CLINICAL TRIAL: NCT05593250
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 2 Study to Evaluate the Efficacy and Safety of SHR-1905 in Subjects With Severe Uncontrolled Asthma.
Brief Title: A Trial of SHR-1905 in Subjects With Severe Uncontrolled Asthma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1905-201
Record Dates: First submitted 2022-10-14; First posted 2022-10-25 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: SHR-1905 compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): dose 1
  Interventions: Drug: SHR-1905
- Cohort B (Experimental): dose 2
  Interventions: Drug: SHR-1905
- Cohort C (Experimental): dose 3
  Interventions: Drug: SHR-1905
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SHR-1905 — subcutaneous
  Arms: Cohort A; Cohort B; Cohort C
Drug: placebo — subcutaneous ,placebo
  Arms: Placebo

SUMMARY:
This study is a phase 2 study of SHR-1905 in subjects with severe uncontrolled asthma. The purpose of the study is to evaluate efficacy and safety of SHR-1905 in subjects with severe uncontrolled asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 75 years (inclusive)
2. Weight ≥ 40 kg
3. Meet the diagnostic criteria for asthma and have a medical history of at least 1 year
4. Treatment with a total daily dose of either medium or high dose inhaled glucocorticoids (ICS) for at least 6 months before screening, with a stable use for 3 months before randomization
5. At least one additional maintenance asthma controller with stable use for at least 3 months before randomization
6. At least 2 exacerbations within 12 months before screening
7. No birth plan and must agree to take effective contraceptive methods
8. Sign informed consent form voluntarily for the trial

Exclusion Criteria:

1. Any clinically important pulmonary disease
2. Any disease other than asthma that may affect lung function
3. Any disease other than asthma related to elevation of eosinophils
4. Any immunodeficiency disease
5. Any clinically important serious cardiovascular diseases unstable or uncontrolled
6. Uncontrolled Hypertension
7. Uncontrolled Diabetes Mellitus
8. Any clinically important infections within 4 weeks before randomization
9. Any major surgery within 3 months before randomized, or any surgical plan during the study, or any treatment that may affect the evaluation of the subjects considered by the investigator
10. Any parasitic infections within 6 months before randomization
11. Malignancy diagnosed within 5 years before randomization
12. Abnormal laboratory tests during screening and baseline
13. Positive infectious disease test
14. Prolonged QTc interval or other clinical significant abnormal findings in ECG at screening that may cause safety risk to the subject
15. Current smoker or smoking cessation for less than 6 months at screening, or smoking history ≥10 pack- years
16. Drug or alcohol abuse
17. Allergy history to any biologicsl or other agent that investigator think the subject should not participate in the study
18. Subjects who are pregnant or breastfeeding, or plan to become pregnant during the study
19. Participated in other clinical trials and used investigational drugs containing active ingredients within 4 weeks or 5 half-lives before screening
20. Any other circumstance inappropriate for participating in the clinical trial considered by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy：Annual asthma exacerbation rate (AAER) | From randomisation to 48 weeks

SECONDARY OUTCOMES:
Changes of fractional exhaled nitric oxide (FeNO) compared with baseline | Baseline to72 weeks
Changes from baseline in Asthma Control questionnaire (ACQ-6) scores | Baseline to 72 weeks
Changes from baseline in Asthmatic Quality of Life Questionnaire (AQLQ) scores | Baseline to 72 weeks
AAER associated with hospitalization at 48 weeks | From randomisation to 48 weeks
Changes from baseline in Asthma Symptom Diary scores | Baseline to 72 weeks
The proportion of subjects with acute exacerbations of asthma | Baseline to 72 weeks
Changes from baseline in weekly reliever use | Baseline to 72 weeks
Changes from baseline in weekly mean morning and evening peak expiratory flow (PEF) | Baseline to 72 weeks
Changes from baseline in weekly mean number of night time awakenings | Baseline to 72 weeks
Time to the first acute asthma exacerbation | Baseline to 72 weeks
The proportion of subjects with composite endpoint for asthma (CompEx) | Baseline to72 weeks
Pharmacokinetics (PK): Serum concentration of SHR-1905 | 72 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided